CLINICAL TRIAL: NCT04502758
Title: A Randomized Controlled Trial of Sequential Bilateral Accelerated Theta Burst Stimulation in Adolescents With Suicidal Ideation Associated With Major Depressive Disorder
Brief Title: Sequential Bilateral Accelerated Theta Burst Stimulation in Adolescents With Suicidal Ideation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Paul E. Croarkin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-009630-1; R01MH124655-01 (NIH); NCT04701840 (obsolete NCT alias)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Suicidal Ideation; Major Depressive Disorder
Keywords: Adolescent
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The use of the MagVenture Cool-B70 A/P coils facilitates blinding of the operator and subjects receiving aTBS or sham treatments. The study team members completing clinical rating scales will also not be allowed in the treatment suite during TBS treatment sessions and will be blinded to treatment assignment. A pre-post treatment expectancy and experience form will ask subjects and parents to make a guess regarding treatment arm (active or sham). Blinded study team members will also be asked to guess treatment assignments for each subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sequential bilateral accelerated theta burst stimulation (Active Comparator): Three sessions of Sequential bilateral accelerated theta burst stimulation (aTBS) are administered daily for 10 days (5 days per week).
  Interventions: Device: MagVenture TMS Therapy System w/Theta Burst Stimulation
- Sham seqential billateral accelerated theta burst stimulation (Sham Comparator): Three sessions of Sequential bilateral sham accelerated theta burst stimulation (aTBS) are administered daily for 10 days (5 days per week).
  Interventions: Device: Sham MagVenture TMS Therapy System w/Theta Burst Stimulation

INTERVENTIONS:
Device: MagVenture TMS Therapy System w/Theta Burst Stimulation — During each session continuous theta burst stimulation (cTBS) in which 1800 pulses are delivered continuously over 120 seconds to the right dorsolateral prefrontal cortex (RDPFC) is administered first, followed by iTBS in which 1800 pulses are delivered in 2 second bursts, repeated every 10 seconds for 570 seconds (1800 pulses) to the left dorsolateral prefrontal cortex (LDPFC). The device consists of a magnetic stimulator, MagPro X100 and a magnetic coil used for MT determination, C-B70 and a treatment coil, the Cool-B70 A/P coil. The A/P version of the coil, contains both an active site (A) and a sham (P) site. The magnetic field properties on the active site are identical to that of the standard Cool-B70 coil, cleared for iTBS treatment.
  Other Names: The MagVenture TMS Therapy System w/Theta Burst Stimulation
  Arms: Sequential bilateral accelerated theta burst stimulation
Device: Sham MagVenture TMS Therapy System w/Theta Burst Stimulation — During each session continuous theta burst stimulation (cTBS) in which 1800 pulses are delivered continuously over 120 seconds to the right dorsolateral prefrontal cortex (RDPFC) is administered first, followed by iTBS in which 1800 pulses are delivered in 2 second bursts, repeated every 10 seconds for 570 seconds (1800 pulses) to the left dorsolateral prefrontal cortex (LDPFC). The device consists of a magnetic stimulator, MagPro X100 and a magnetic coil used for MT determination, C-B70 and a treatment coil, the Cool-B70 A/P coil. The A/P version of the coil, contains both an active site (A) and a sham (P) site. The magnetic field on the sham site is significantly reduced, and is less than 5% of that of the active site.
  Arms: Sham seqential billateral accelerated theta burst stimulation

SUMMARY:
The purpose of this study is to gather information regarding the use of a new type of transcranial magnetic stimulation (TMS) called theta burst stimulation (TBS) for suicidal ideation in adolescents with Major Depressive Disorder (MDD). The investigators hope to learn if this TMS treatment improves suicidal ideation over 10 days and clinical outcomes over 1 year of follow-up.

DETAILED DESCRIPTION:
The proposed study will examine sequential bilateral accelerated theta burst stimulation (aTBS). Three sessions are administered daily for 10 days (5 days per week). During each session continuous theta burst stimulation (cTBS) in which 1800 pulses are delivered continuously over 120 seconds to the right dorsolateral prefrontal cortex (RDPFC) is administered first, followed by iTBS in which 1800 pulses are delivered in 2 second bursts, repeated every 10 seconds for 570 seconds (1800 pulses) to the left dorsolateral prefrontal cortex (LDPFC). The theta burst stimulation (TBS) parameters were adopted from prior work, with 3-pulse 50 Hz bursts given every 200 ms (at 5 Hz) with an intensity of 80% of active motor threshold. The comparison group will receive 3 daily sessions of bilateral sham TBS treatment for 10 days. Subjects in both groups will take part in a daily psychotherapeutic treatment program.

The proposed study will examine sequential bilateral accelerated theta burst stimulation (aTBS). Three sessions are administered daily for 10 days (5 days per week). During each session continuous theta burst stimulation (cTBS) in which 1800 pulses are delivered continuously over 120 seconds to the right dorsolateral prefrontal cortex (RDPFC) is administered first, followed by iTBS in which 1800 pulses are delivered in 2 second bursts, repeated every 10 seconds for 570 seconds (1800 pulses) to the left dorsolateral prefrontal cortex (LDPFC). The theta burst stimulation (TBS) parameters were adopted from prior work, with 3-pulse 50 Hz bursts given every 200 ms (at 5 Hz) with an intensity of 80% of active motor threshold. The comparison group will receive 3 daily sessions of bilateral sham TBS treatment for 10 days. Subjects in both groups will take part in a daily psychotherapeutic treatment program.

The study will enroll outpatient and inpatient adolescents (aged 12-18 years) with Major Depressive Disorder (MDD) of at least moderate severity defined as a Children's Depression Rating Scale Revised (CDRS-R) Score of 40 or greater and suicidal ideation defined as a score of 3 or greater on item 13 (Suicidal Ideation) of the CDRS-R.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients
* Voluntary clinical patient with the capacity to assent to treatment and a parent or legal guardian with the capacity to consent
* Female or male
* 12-18 years of age
* Diagnosed with MDD based on Diagnostic and Statistical Manual for Mental Disorders, 5th edition (DSM-5) criteria122 with the Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI Kid) in subjects 12-17 years of age;118 The Mini-International Neuropsychiatric Interview will be used for subjects who are 18 years of age117
* In a current episode of MDD with duration of at least 4 weeks but less than 3 years
* Depressive symptom severity as demonstrated by CDRS-R total composite score of 40 or greater and a suicidal ideation score of 3 or more on item 13 of the CDRS-R109
* Demonstrating that depressive symptom severity as evaluated at the screening visit does not improve between screening and baseline by 25% or more
* Eligible for transcranial magnetic stimulation (TMS) based on safety criteria104
* On a medically acceptable form of birth control if female
* Taking an antidepressant medication if recommended by the referring clinician and agreed upon by parents and patients. Please note that patients are not required to take an antidepressant medication for study participation for practical, ethical, and human subject protection concerns. Medication status and prior treatment resistance will be carefully recorded with the Antidepressant Treatment History Form113 criteria for relevant statistical considerations.

Exclusion Criteria:

* Diagnosis of a psychotic disorder, bipolar disorder, anorexia nervosa, bulimia nervosa, substance use disorders within the past year (with the exception of caffeine and tobacco).
* Intelligent quotient less than 70 (if there is a clinical concern, subjects will be psychometrically assessed with the Slosson Intelligence Test, Revised).123
* Positive urine drug screen at baseline
* Seizure history
* Any family history of epilepsy
* History of any treatment with electroconvulsive therapy or TMS
* Use of any investigational drug within 4 weeks of baseline
* Prior brain surgery
* Risk for increased intracranial pressure such as a brain tumor
* Head trauma with loss of consciousness
* Any true positive findings on the TMS safety screening form
* Pregnancy or suspected pregnancy
* Conductive, ferromagnetic, or other magnetic-sensitive metals implanted in the head-within 30 cm of the treatment coil excluding the mouth that cannot be safely removed (examples include cochlear implants, vagus nerve stimulators, deep brain stimulators, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes).
* Implanted medication pumps and cardiac pacemakers
* Any unstable medical condition
* Inability to adhere to the protocol

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | up to 12 months
  Suicidal Ideation as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS). This is a validated, clinician-rated tool collected to assess lifetime and ongoing suicidal ideation and behavior. The severity of ideation subscale is a 5-point ordinal scale 1-5 . 1 = Wish to be dead - 5 = Active Suicidal Ideation with Specific Plan and Intent. Assessed at baseline, 10 days and 12 months.
Hospitalizations | up to 12 months
  The total number of hospitalizations related to suicide idealization

SECONDARY OUTCOMES:
Cortical inhibition | baseline, 10 days
  As measured in Changes in test stimulus (TS) motor evoked potential (MEP) amplitude of are expressed as a percentage of the mean unconditioned MEP amplitude. For N100 response data collection, mean single pulse data will be collected for each electrode for the TMS-evoked potential. The N100 peak value is then extracted throughout electrodes from the negative in closest proximity to 100 ms.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Croarkin, DO, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded and NIMH databases and shared as per NIMH and NIH policy

REFERENCES:
- [Background] Sonmez AI, Camsari DD, Nandakumar AL, Voort JLV, Kung S, Lewis CP, Croarkin PE. Accelerated TMS for Depression: A systematic review and meta-analysis. Psychiatry Res. 2019 Mar;273:770-781. doi: 10.1016/j.psychres.2018.12.041. Epub 2018 Dec 7. PMID 31207865
- [Background] Lewis CP, Camsari DD, Sonmez AI, Nandakumar AL, Gresbrink MA, Daskalakis ZJ, Croarkin PE. Preliminary evidence of an association between increased cortical inhibition and reduced suicidal ideation in adolescents treated for major depression. J Affect Disord. 2019 Feb 1;244:21-24. doi: 10.1016/j.jad.2018.09.079. Epub 2018 Sep 28. PMID 30292987
- [Background] Croarkin PE, Nakonezny PA, Deng ZD, Romanowicz M, Voort JLV, Camsari DD, Schak KM, Port JD, Lewis CP. High-frequency repetitive TMS for suicidal ideation in adolescents with depression. J Affect Disord. 2018 Oct 15;239:282-290. doi: 10.1016/j.jad.2018.06.048. Epub 2018 Jul 18. PMID 30031247
- [Background] Lewis CP, Nakonezny PA, Blacker CJ, Vande Voort JL, Port JD, Worrell GA, Jo HJ, Daskalakis ZJ, Croarkin PE. Cortical inhibitory markers of lifetime suicidal behavior in depressed adolescents. Neuropsychopharmacology. 2018 Aug;43(9):1822-1831. doi: 10.1038/s41386-018-0040-x. Epub 2018 Mar 14. PMID 29703993
- [Background] Dhami P, Knyahnytska Y, Atluri S, Lee J, Courtney DB, Croarkin PE, Blumberger DM, Daskalakis ZJ, Farzan F. Feasibility and clinical effects of theta burst stimulation in youth with major depressive disorders: An open-label trial. J Affect Disord. 2019 Nov 1;258:66-73. doi: 10.1016/j.jad.2019.07.084. Epub 2019 Jul 30. PMID 31398593
- [Derived] Yuruk D, Ozger C, Garzon JF, Leffler JM, Shekunov J, Vande Voort JL, Zaccariello MJ, Nakonezny PA, Croarkin PE. Sequential bilateral accelerated theta burst stimulation in adolescents with suicidal ideation associated with major depressive disorder: Protocol for a randomized controlled trial. PLoS One. 2023 Apr 13;18(4):e0280010. doi: 10.1371/journal.pone.0280010. eCollection 2023. PMID 37053246
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials